CLINICAL TRIAL: NCT06342856
Title: Evaluation of Treatment With Coenzyme Q10 and L-Carnitine on Semen Parameters in Infertile Men With Idiopathic Oligoasthenoteratospermia a Placebo Controlled Clinical Trial
Brief Title: Evaluation of Treatment With Coenzyme Q10 and L-Carnitine on Semen Parameters in Infertile Men With Idiopathic Oligoasthenoteratospermia
Acronym: infertility
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: idiopathic infertility
Record Dates: First submitted 2024-03-08; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2023-08

CONDITIONS: Infertility Unexplained; Oligospermia
Keywords: infertility; oligospermia; coenzyme Q1o
MeSH Terms: conditions — Oligospermia; Infertility | interventions — Ubiquinone; Carnitine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): will receive a daily dose of 200 mg of CoQ10 for 3 months
  Interventions: Drug: co enzyme Q10 , L- Carnitine
- Group 2 (Active Comparator): will receive L-carnitine 1 tablet per day orally for 3 months
  Interventions: Drug: co enzyme Q10 , L- Carnitine
- Group 3 (Active Comparator): will receive combination of a daily dose of 200 mg of CoQ10 and 1 tablet of L-carnitine for 3 months
  Interventions: Drug: co enzyme Q10 , L- Carnitine
- Group 4 (Placebo Comparator): will receive a placebo for 3 months
  Interventions: Drug: co enzyme Q10 , L- Carnitine

INTERVENTIONS:
Drug: co enzyme Q10 , L- Carnitine — Patient fulfilling inclusion criteria after obtaining consent will be randomized into four equal groups randomization will be computer based

SUMMARY:
Evaluation of treatment with Coenzyme Q10 and L-Carnitine on Semen Parameters in Infertile men with Idiopathic Oligoasthenoteratospermia

DETAILED DESCRIPTION:
Evaluation of treatment with Coenzyme Q10 and L-Carnitine on Semen Parameters in Infertile men with Idiopathic Oligoasthenoteratospermia a placebo controlled clinical trial

ELIGIBILITY:
Inclusion Criteria:

* of in¬fertility of 1 year or more without the use of contraception

Exclusion Criteria:

* o Active genital infections.

  * Patients with ejaculatory dysfunction
  * Azoospermia

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — semen analysis
Enrollment: 120 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Semen analysis parameters compared to baseline | 6 months
  Changes in Semen analysis parameters compared to baseline

SECONDARY OUTCOMES:
Serum hormone levels ([FSH], [LH], testosterone, and prolactin) levels compared to baseline and Cost analysis | 6 moths
  Serum hormone levels ([FSH], [LH], testosterone, and prolactin) levels compared to baseline and Cost analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Result] Salvio G, Cutini M, Ciarloni A, Giovannini L, Perrone M, Balercia G. Coenzyme Q10 and Male Infertility: A Systematic Review. Antioxidants (Basel). 2021 May 30;10(6):874. doi: 10.3390/antiox10060874. PMID 34070761